CLINICAL TRIAL: NCT07133399
Title: Relative Bioavailability of Two Different Vicadrostat/ Empagliflozin Combinations and Investigation of the Effect of Food on the Pharmacokinetics of a Vicadrostat/ Empagliflozin Combination in Healthy Male and Female Volunteers (an Open-label, Randomised, Single-dose, Three- Way Crossover Study)
Brief Title: A Study in Healthy People to Test How 2 Different Formulations of a Combination Treatment (Vicadrostat and Empagliflozin) Are Taken up in the Body and How Food Influences the Amount of the Medicines in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1378-0043; 2025-521650-42-00 (Registry Identifier: CTIS); U1111-1319-1746 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-08-19; First posted 2025-08-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: three-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R -T1 -T2 (Experimental): R = reference (vicadrostat / empagliflozin combination 1) fasted T1 = test 1 (vicadrostat / empagliflozin 2) fasted T2 = test 2 (vicadrostat / empagliflozin 1) fed
  Interventions: Drug: vicadrostat / empagliflozin combination 1; Drug: vicadrostat / empagliflozin 2
- T1 - R - T2 (Experimental): R = reference (vicadrostat / empagliflozin combination 1) fasted T1 = test 1 (vicadrostat / empagliflozin 2) fasted T2 = test 2 (vicadrostat / empagliflozin 1) fed
  Interventions: Drug: vicadrostat / empagliflozin combination 1; Drug: vicadrostat / empagliflozin 2

INTERVENTIONS:
Drug: vicadrostat / empagliflozin combination 1 — vicadrostat / empagliflozin combination 1
Drug: vicadrostat / empagliflozin 2 — vicadrostat / empagliflozin 2

SUMMARY:
To investigate the relative bioavailability of two different vicadrostat/empagliflozin combinations. Additionally, the trial investigates the effect of food on the pharmacokinetics of the vicadrostat/empagliflozin.

ELIGIBILITY:
Inclusion Criteria :

1. Healthy male or female trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body Mass Index (BMI) of 18.5 to 29.9 kg / m^2 (inclusive)
4. Signed and dated written informed consent in accordance with Harmonized Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. For female trial participants: Female trial participants who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
   * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) plus condom
   * Sexually abstinent (if refraining from heterosexual intercourse is the preferred and usual lifestyle of the subject).
   * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
   * Surgically sterilised (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal ligation)
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause.

Exclusion Criteria:

1. Any finding in the medical examination (including Blood pressure (BP) Pulse rate (PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 105 to 140 mmHg, diastolic blood pressure outside the range of 65 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | Up to 4 days
Maximum measured concentration of the analyte in plasma (C max) | Up to 4 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞) | Up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com